CLINICAL TRIAL: NCT05786560
Title: BABE(Body Appreciation and Better Eating), Add Some Self-compassion: a Randomized Controlled Pilot Study for Black/African American High School Teenage Girls
Brief Title: BABE(Body Appreciation and Better Eating), Add Some Self-compassion
Acronym: BABE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Nkechi Okpara, Principal Investigator, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00120545
Record Dates: First submitted 2022-12-29; First posted 2023-03-27 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Body Image; Eating Behavior; Binge Eating; Nutrition, Healthy; Disordered Eating
MeSH Terms: conditions — Feeding Behavior; Bulimia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body image + nutrition education +self-compassion (Experimental): For the treatment arm, girls will participate in the Body Project for about 30 minutes, then will be given about a 30 minute self-compassion-based nutrition education lesson. The nutrition topics will cover the basic biochemistry of nutrition, nutrition needs for teenage girls, and ways to find balance in eating, framed in the constructs of self-compassion. The three self-compassion constructs will be targeted in the following ways: (1) Mindfulness will involve bringing awareness to feelings and emotions about a time during the week where participants ate a food lower in nutritional value. (2) Common Humanity involves finding ways in which their experience connects to others and acknowledging that being human comes with imperfections. (3) Self-Kindness will involve having girls speak kind and understanding words to themselves as it relates to their eating-related downfall of the week.
  Interventions: Behavioral: BABE (Body Appreciation and Better Eating)
- Body image + nutrition education (Active Comparator): For the control arm, participants will receive the same 30-minute Body Project class, then participants will be given a 30-minute nutrition education lesson. The nutrition lesson plans will have no components of self-compassion intertwined within the lesson, but the nutrition content will be the same as the treatment group.
  Interventions: Behavioral: BABE (Body Appreciation and Better Eating)

INTERVENTIONS:
Behavioral: BABE (Body Appreciation and Better Eating) — The participants will be randomized into either a treatment or control group. For the treatment arm, girls will participate in the Body Project for 30 minutes, then will be given a 30-minute self-compassion-based nutrition education lesson. Nutrition topics will cover the basic biochemistry of nutrition, nutrition needs for teenage girls, and ways to find balance in eating, framed in the constructs of self-compassion. The control group will receive the same 30-minute Body Project class and the same 30-minute nutrition education class; however, there will be no incorporation of self-compassion.

SUMMARY:
Body dissatisfaction is most common among girls in their teenage years and young adulthood, this is also around the time where the risk of developing binge eating disorder is the highest. Black/African American girls are more likely to engage in binge eating behaviors compared to their White American counterparts; however, they receive less help for eating issues. Further, increase rates of obesity in the Black/African American population may indicate that binge eating may be a bigger problem for this population than discussed. Therefore, the primary purpose of this randomized controlled pilot is to assess the feasibility of this pilot study to be used in a large scale fully-powered study. The secondary purpose of this study is to assess if two different nutrition and body image programs elicit positive outcomes among Black/African American teenage girls who indicate a desire to improve body image.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Black (Afro-Latina)/African American teenage girls
* Age 13 to 18 years old
* Attend high school in the United States
* Interest in nutrition

Exclusion Criteria:

* Eating disorder diagnosis
* Pregnancy

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the BABE program (sample size) | 12 weeks
  The feasibility of this randomized controlled pilot will consider sample size. Feasibility will be measured by the length of time required to complete participant recruitment (=20-24).
Feasibility of the BABE program (retention) | 12 weeks
  The feasibility of this randomized controlled pilot will consider retention. Feasibility will be measured by the retention rate/response rate (100 %) at 1-month follow-up.
Feasibility of the BABE program (randomization) | 12 weeks
  The feasibility of this randomized controlled pilot will consider randomization. Feasibility will be measured by the ability to randomize participants (if researcher needs to add additional class options to accommodate teen girls).
Participants' acceptability of the program | 12 weeks
  Program acceptability will be measured by focus groups conducted post-intervention and a credibility scale which will be given after classes. The Credibility scale measures the degree to which participants believe their intervention is credible and effective in improving outcomes (body image and nutrition). Some of the question items included, "How logical is this program in helping you improving eating habits? How logical is this program in helping you improve body image? Responses are indicated on a 9-point Likert scale of 0 (not at all) to 9 (very). Higher scores mean better outcomes.

SECONDARY OUTCOMES:
Self-compassion for youth scale | 12 weeks
  My secondary objectives will test within and between groups (treatment vs control) changes in self-compassion. The Self-Compassion Scale for youth consists of 17 items to assess self-compassion through the components of self-kindness, self-judgment. Responses are indicated on a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Higher scores mean better outcomes.
Body Appreciation Scale-2 | 12 weeks
  My secondary objectives will test within and between groups (treatment vs control) changes in body appreciation. The Body appreciation scale-2 (BAS-2) consists of 10 items that measure body appreciation by assessing individuals' acceptance of favorable opinions towards and respect for their bodies. Responses are indicated on a 5-point Likert scale from 1 (never) to 5 (always). Higher scores mean better outcomes.
Mindful eating questionnaire | 12 weeks
  My secondary objectives will test within and between groups (treatment vs control) changes in mindful eating. The Mindful Eating Questionnaire for Children (MEQ-C) is a 17-item questionnaire that consists of five subscales: disinhibition, awareness, external cues, emotional response, and distraction. Responses are indicated on a Likert scale from 1 (never/rarely) to 4 (usually/always), with higher scores indicating greater degrees of mindful eating.
Childrens Brief Binge Eating Questionnaire | 12 weeks
  My secondary objectives will test within and between groups (treatment vs control) changes in binge eating. The Children's Brief Binge-Eating Questionnaire (CBBEQ) consists of 7 questions and responses are provided on a Likert-type scale from "Definitely false" (0) to "Definitely true" (3). Higher scores mean greater risk for binge eating disorder.
Motivations for Electronic Interaction Scale (MEIS) | 12 weeks
  My secondary objectives will test within and between groups (treatment vs control) changes in motivation for using social media. The Motivations for Electronic Interaction Scale (MEIS) assesses adolescents' attitudes and behaviors regarding the use of "electronic interaction." The social comparison and feedback-seeking subscale is a 10-item measure, assessing adolescents' use of social media to "seek out information regarding one's appearance, behaviors, and social status, relative to one's peers. Responses are indicated on a 5-point Likert scale (1 for Not at all true, and 5 for Extremely true). Higher scores mean worse outcomes.
The Social Connectedness Scale | 12 weeks
  My secondary objectives will test within and between groups (treatment vs control) changes in social connectedness. The Social Connectedness Scale (SCS) assesses the degree to which youth feel connected to others in their social environment. The SCS is an eight-item measure. Responses are indicated on a six-point Likert scale ranging from 1 (agree) to 6 (disagree). Higher scores mean better outcomes.
Body-Related Shame and Guilt Scale (WEB-SG) | 12 weeks
  My secondary objectives will test within and between groups (treatment vs control) changes in eating guilt. The WEB-SG is a 12-item scale that measures feelings of shame (six items) and guilt (six items). This study will only utilize the guilt scale. Responses will be indicated on a 5-point scale from 0 "never" to 4 "always." Higher scores mean worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nkechi Okpara, MS, RDN, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol